CLINICAL TRIAL: NCT04236310
Title: A Study of Neoadjuvant SHR6390 in Combination With Anastrozole, Pyrotinib, and Trastuzumab in Patients With ER-Positive, HER2-Positive Breast Cancer.
Brief Title: A Study of Neoadjuvant SHR6390 in Combination With Anastrozole, Pyrotinib, and Trastuzumab in Patients With ER+/HER2+ Breast Cancer.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJBC2001
Record Dates: First submitted 2020-01-17; First posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Breast Cancer; HER2-positive Breast Cancer; ER-positive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; pyrotinib; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR6390+Anastrozole+Pyrotinib+Trastuzumab±Ovarian Suppression (Experimental)
  Interventions: Drug: SHR6390; Drug: Anastrozole; Drug: Pyrotinib; Drug: Trastuzumab

INTERVENTIONS:
Drug: SHR6390 — SHR6390 150 mg, orally once daily on Day 1 to Day 21 of every 28-day cycle followed by 7 days off treatment for 4 cycles
Drug: Anastrozole — Anastrozole 1md, orally once daily for 16 weeks (For premenopausal women, ovarian suppression may be considered)
Drug: Pyrotinib — Pyrotinib 400mg once daily for 16 weeks
Drug: Trastuzumab — Trastuzumab 6mg/kg (loading dose, 8mg/kg), infusion once every 3-week cycle for 5 cycles.

SUMMARY:
To evaluate the efficacy and safety of the SHR6390 in combination with anastrozole, pyrotinib, and trastuzumab in patients with ER-positive, HER2-positive breast cancer in the neoadjuvant setting.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent for all study according to local regulatory requirements prior to beginning specific protocol procedures.
2. Age at diagnosis ≥18 years and ≤75 years, female.
3. Histologically confirmed diagnosis of Unilateral ER+/HER2+ breast cancer. ER-positivity is defined as >1% stained cells；HER2-positivity is defined as IHC 3+ or if IHC scored 2+, in-situ hybridisation (ISH) suggests amplified HER2 gene.
4. Tumor diameter >2 centimeters with the clinical stage being classified as from IIa to IIIc.
5. ECOG ≤ 1, LVEF ≥ 55%.
6. Laboratory requirements: for hematology, absolute neutrophil count (ANC) ≥1.5 × 109 / L and platelets ≥100 × 109 / L and hemoglobin ≥90 g/L; for hepatic function, total bilirubin ≤1.5 × UNL, AST and ALT ≤2.5 × UNL; for renal function, SCr ≤1.5 × UNL.

Exclusion Criteria:

1. Evidence of bilateral invasive breast cancer or metastatic disease (M1).
2. Pevious treatment with chemotherapy, hormonal therapy, an investigational drug for any type of malignancy, or radiation therapy.
3. Any of the following exist in the last 6 months: known or suspected congestive heart failure (≥ NYHA II), persistent arrhythmias (≥ grade 2), atrial fibrillation of any grade, coronary / peripheral bypass, symptomatic congestive heart failure, cerebrovascular accidents (including transient cerebral hemorrhage attacks or symptomatic pulmonary embolism).
4. Known hypersensitivity reaction to one of the compounds or incorporated substances used in this protocol.
5. Active infection or severe symptomatic visceral disease in the last 4 weeks.
6. Patients with HIV infection or known AIDS, or patients with infection of active hepatitis B (HBV DNA ≥1000IU / ml) or hepatitis C (hepatitis C antibody is positive and HCV RNA is above the lower limit of detection of the analytical method).
7. Prior malignancy with a disease-free survival of < 5 years, except curatively treated basalioma of the skin, pTis of the cervix uteri.
8. Pregnant or lactating patients. Patients of childbearing potential must implement adequate non-hormonal contraceptive measures (barrier methods, intrauterine contraceptive devices, sterilization) during study treatment.
9. Participation in another clinical trial with any investigational, not marketed drug within 30 days prior to study entry.
10. Not eligible for the trial assessed by the investigators of our study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2020-01-15 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Ki67 changes from baseline to 2 weeks after the start of the neoadjuvant therapy | 2 weeks
  Ki67 changes from baseline to at 2 weeks after the start of the neoadjuvant therapy

SECONDARY OUTCOMES:
Ki67 changes from baseline to at surgery | average 19 weeks after the start of the neoadjuvant therapy
  Ki67 changes from baseline to at surgery
Pathological complete response (ypT0/is ypN0) rate | average 19 weeks after the start of the neoadjuvant therapy
  Absence of invasive cancer in the breast and axillary nodes, irrespective of ductal carcinoma in situ.
Objective response rate (ORR) | average 19 weeks after the start of the neoadjuvant therapy
  ORR includes all patients whose cancer has a partial or complete response according to RECIST 1.1
Invasive disease-free survival (IDFS) | 5 years
  IDFS is defined as the time period between registration and first event (ipsilateral invasive breast tumor recurrence, regional invasive breast cancer recurrence, distant recurrence, death attributable to any cause, contralateral invasive breast cancer, second primary nonbreast invasive cancer)
Tolerability and safety: number of patients whose treatment had to be reduced, delayed or permanently stopped | during treatment (16 weeks)
  Descriptive statistics will be given on the number of patients whose treatment had to be reduced, delayed or permanently stopped.

IPD SHARING:
Plan to Share IPD: No